CLINICAL TRIAL: NCT02888743
Title: A Phase 2 Study of MEDI4736 (Durvalumab) and Tremelimumab Alone or in Combination With High or Low-Dose Radiation in Metastatic Colorectal and NSCLC
Brief Title: Durvalumab and Tremelimumab With or Without High or Low-Dose Radiation Therapy in Treating Patients With Metastatic Colorectal or Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2016-01325; NCI-2016-01325 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17-719; 10021 (Other: Dana-Farber - Harvard Cancer Center LAO); 10021 (Other: CTEP); UM1CA186709 (NIH)
Record Dates: First submitted 2016-08-31; First posted 2016-09-05 (Estimated); Results first posted 2024-06-25 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Colorectal Carcinoma; Metastatic Lung Non-Small Cell Carcinoma; Stage IV Colorectal Cancer AJCC v7; Stage IV Lung Non-Small Cell Cancer AJCC v7; Stage IVA Colorectal Cancer AJCC v7; Stage IVB Colorectal Cancer AJCC v7
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; Immunoglobulin G; Disulfides; Radiotherapy; Radiation; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1, Arm A (tremelimumab, durvalumab, HD-RT) (Experimental): Patients receive tremelimumab and durvalumab and as in Arm C. Beginning at week 2, patients receive high dose radiation therapy QD over 10 days for up to 3 fractions.
  Interventions: Biological: Durvalumab; Radiation: Radiation Therapy; Biological: Tremelimumab
- Cohort 1, Arm B (tremelimumab, Durvalumab, LD-RT) (Experimental): Patients receive tremelimumab and durvalumab and as in Arm C. Beginning at week 2, patients receive low dose radiation therapy every 6 hours BID on weeks 2, 6, 10 and 14.
  Interventions: Biological: Durvalumab; Radiation: Radiation Therapy; Biological: Tremelimumab
- Cohort 1, Arm C (tremelimumab, durvalumab) (Experimental): Patients receive tremelimumab IV and durvalumab IV over 60 minutes every 4 weeks for up to 16 weeks in the absence of disease progression or unacceptable toxicity. Patients then receive durvalumab IV over 60 minutes 4 weeks after last combination dose for up to 9 additional doses.
  Interventions: Biological: Durvalumab; Biological: Tremelimumab
- Cohort 2, Arm A (tremelimumab, durvalumab, HD-RT) (Experimental): Patients receive tremelimumab IV and durvalumab IV over 60 minutes every 4 weeks for up to 16 weeks in the absence of disease progression or unacceptable toxicity. Patients then receive durvalumab IV over 60 minutes 4 weeks after last combination dose for up to 9 additional doses. Beginning at week 2, patients receive high dose radiation therapy QD over 10 days for up to 3 fractions.
  Interventions: Biological: Durvalumab; Radiation: Radiation Therapy; Biological: Tremelimumab
- Cohort 2, Arm B (tremelimumab, durvalumab, LD-RT) (Experimental): Patients receive tremelimumab IV and durvalumab IV over 60 minutes every 4 weeks for up to 16 weeks in the absence of disease progression or unacceptable toxicity. Patients then receive durvalumab IV over 60 minutes 4 weeks after last combination dose for up to 9 additional doses. Beginning at week 2, patients receive low dose radiation therapy every 6 hours BID on weeks 2, 6, 10 and 14.
  Interventions: Biological: Durvalumab; Radiation: Radiation Therapy; Biological: Tremelimumab

INTERVENTIONS:
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI 4736; MEDI-4736; MEDI4736
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: Cohort 1, Arm A (tremelimumab, durvalumab, HD-RT); Cohort 1, Arm B (tremelimumab, Durvalumab, LD-RT); Cohort 2, Arm A (tremelimumab, durvalumab, HD-RT); Cohort 2, Arm B (tremelimumab, durvalumab, LD-RT)
Biological: Tremelimumab — Given IV
  Other Names: Anti-CTLA4 Human Monoclonal Antibody CP-675,206; CP 675; CP 675206; CP-675; CP-675,206; CP-675206; CP675; CP675206; Imjudo; Ticilimumab; Tremelimumab-actl

SUMMARY:
This randomized phase II trial studies the side effects of durvalumab and tremelimumab and to see how well they work with or without high or low-dose radiation therapy in treating patients with colorectal or non-small cell lung cancer that has spread to other parts of the body (metastatic). Immunotherapy with durvalumab and tremelimumab, may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Giving durvalumab and tremelimumab with radiation therapy may work better in treating patients with colorectal or non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess safety and tolerability of combined checkpoint blockade with MEDI4736 (durvalumab) and tremelimumab alone or with high or low-dose radiation in non-small cell lung cancer (NSCLC). (NSCLC Cohort) II. To compare the overall response (excluding the irradiated lesion[s]) between combined checkpoint blockade with MEDI4736 and tremelimumab alone or combined checkpoint blockade with low or high dose radiation. (NSCLC Cohort) III. To assess safety and tolerability of combined checkpoint blockade with MEDI4736 and tremelimumab with high or low-dose radiation. (Colorectal Cohort) IV. To determine the overall response rate (excluding the irradiated lesion[s]) with combined checkpoint blockade with MEDI4736 and tremelimumab with either low or high dose radiation. (Colorectal Cohort)

SECONDARY OBJECTIVES:

I. To estimate median progression-free survival and overall survival. (NSCLC Cohort) II. To determine local control within the irradiated field(s) and abscopal response rates. (NSCLC Cohort) III. To evaluate associations between PD-L1 expression as well as levels of infiltrating CD3+, CD8+ T-cells and overall response. (NSCLC Cohort) IV. To explore changes in PD-L1 expression, circulating T-cell populations, T-cell infiltration, ribonucleic acid (RNA) expression, spatial relationship of immune markers, and mutational burden as a result of low or high dose radiation. (NSCLC Cohort) V. To estimate median progression-free survival and overall survival. (Colorectal Cohort) VI. To determine local control within the irradiated field and abscopal response rates. (Colorectal Cohort) VII. To evaluate associations between PD-L1 expression as well as levels of infiltrating CD3+ CD8+ T-cells and overall response. (Colorectal Cohort) VIII. To evaluate changes between PD-L1 expression as well as levels of infiltrating CD3+, CD8+ T-cells induced by targeted low or high dose radiation. (Colorectal Cohort) IX. To explore changes in circulating T-cell populations, T-cell infiltration, RNA expression, spatial relationship of immune markers, and mutational burden as a result of low or high dose radiation. (Colorectal Cohort)

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT 1: Patients with NSCLC are randomized to 1 of 3 arms.

ARM A: Patients receive tremelimumab and durvalumab and as in Arm C. Beginning at week 2, patients receive high dose radiation therapy once per day (QD) over 10 days for up to 3 fractions.

ARM B: Patients receive tremelimumab and durvalumab and as in Arm C. Beginning at week 2, patients receive low dose radiation therapy every 6 hours twice per day (BID) on weeks 2, 6, 10 and 14.

ARM C: Patients receive tremelimumab intravenously (IV) and durvalumab IV over 60 minutes every 4 weeks for up to 16 weeks in the absence of disease progression or unacceptable toxicity. Patients then receive durvalumab IV over 60 minutes 4 weeks after last combination dose for up to 9 additional doses.

COHORT 2: Patients with CRC are randomized to 1 of 2 arms.

ARM A: Patients receive tremelimumab intravenously (IV) and durvalumab IV over 60 minutes every 4 weeks for up to 16 weeks in the absence of disease progression or unacceptable toxicity. Patients then receive durvalumab IV over 60 minutes 4 weeks after last combination dose for up to 9 additional doses. Beginning at week 2, patients receive high dose radiation therapy once per day (QD) over 10 days for up to 3 fractions.

ARM B: Patients receive tremelimumab intravenously (IV) and durvalumab IV over 60 minutes every 4 weeks for up to 16 weeks in the absence of disease progression or unacceptable toxicity. Patients then receive durvalumab IV over 60 minutes 4 weeks after last combination dose for up to 9 additional doses. Beginning at week 2, patients receive low dose radiation therapy every 6 hours twice per day (BID) on weeks 2, 6, 10 and 14.

After completion of study treatment, patients are followed for up to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed non-small cell lung cancer (cohort 1) or colorectal cancer (cohort 2)
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm (>= 2 cm) with conventional techniques or as >= 10 mm (>= 1.5 cm) with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* Patients in both cohorts must have progressive disease following prior therapy; specifically:

  * Cohort 1 (NSCLC): Patients must have evidence of radiologic or clinical disease progression during previous treatment with systemic PD-1 directed therapy and/or have been deemed not to derive clinical benefit from PD-1 directed treatment; this includes patients who demonstrated an initial response and subsequent progression; no prior treatment with chemotherapy or targeted agents are required; intervening therapy is allowed between previous PD-1 directed treatment and there is no required interval from prior PD-1 treatment required; PD-1 directed treatment includes treatment with antibodies targeting the PD-1 receptor such as pembrolizumab or nivolumab, as well as PD-L1 targeted antibodies such as MEDI4736 (durvalumab), atezolizumab and avelumab; these agents may have been administered as part of a clinical trial
  * Cohort 2 (colorectal cancer): Patients must have progressed on >= one-line chemotherapy
* At least 21 days must have elapsed from prior systemic therapy (chemotherapy or radiation)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 60%) and life expectancy greater than 6 months; furthermore, enrollment of patients with greater than 10 measurable lesions is discouraged
* Patients must have normal organ and marrow function independent of transfusion for at least 7 days prior to screening and independent of growth factor support for at least 14 days prior to screening
* Hemoglobin (Hgb) >= 9 g/dl
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 x normal institutional limits; this will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia [predominantly unconjugated bilirubin] in the absence of evidence of hemolysis or hepatic pathology), who will be allowed in consultation with their physician
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) = < 2.5 x institutional upper limit of normal; for patients with hepatic metastases, ALT and AST =< 5 x ULT
* Measured creatinine clearance (CL) > 40 mL/min OR calculated creatinine clearance (CL) > 40 mL/min as determined by Cockcroft-Gault (using actual body weight)
* Patients must have at least one lesion that has not previously been irradiated (and is not within a previously radiated field) and for which palliative radiation is potentially indicated and could be safely delivered at the radiation doses specified in this protocol; this lesion must not be the only measurable lesion so that it is still possible to determine the response rate outside of the radiation treatment field; this lesion must not be within the central nervous system (CNS) (brain or spinal cord) or requiring urgent or emergent palliative radiation given the timing of radiation specified on this protocol; furthermore, this lesion:

  * For cohort 1 (NSCLC cohort) - the lesion to be irradiated must be in the lung, lymph nodes, adrenal gland or liver
  * For cohort 2 (colorectal cohort) - the lesion to be irradiated must be in the liver
* The effects of MEDI4736 and tremelimumab on the developing human fetus are unknown; for this reason and because radiation is known to be teratogenic, evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients is required; women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause; the following age-specific requirements apply:

  * Women < 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy)
  * Women >= 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced oophorectomy with last menses > 1 year ago, had chemotherapy-induced menopause with > 1 year interval since last menses, or underwent surgical sterilization (bilateral oophorectomy or hysterectomy)
* Females of childbearing potential who are sexually active with a non sterilized male partner must use at least 1 highly effective method of contraception from the time of screening and must agree to continue using such precautions for 180 days after the last dose of durvalumab + tremelimumab combination therapy or 90 days after the last dose of durvalumab monotherapy; non-sterilized male partners of a female patient must use male condom plus spermicide throughout this period; cessation of birth control after this point should be discussed with a responsible physician; not engaging in sexual activity for the total duration of the drug treatment and the drug washout period is an acceptable practice; however, periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control; female patients should also refrain from breastfeeding throughout this period
* Non-sterilized males who are sexually active with a female partner of childbearing potential must use a male condom plus spermicide from screening through 180 days after receipt of the final dose of durvalumab + tremelimumab combination therapy or 90 days after receipt of the final dose of durvalumab monotherapy; not engaging in sexual activity is an acceptable practice; however, occasional abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception; male patients should refrain from sperm donation throughout this period
* Female partners (of childbearing potential) of male patients must also use a highly effective method of contraception throughout this period
* Highly effective methods of contraception, defined as one that results in a low failure rate (ie, less than 1% per year) when used consistently and correctly are described in the table below; note that some contraception methods are not considered highly effective (e.g. male or female condom with or without spermicide; female cap, diaphragm, or sponge with or without spermicide; non-copper containing intrauterine device; progestogen-only oral hormonal contraceptive pills where inhibition of ovulation is not the primary mode of action [excluding Cerazette/desogestrel which is considered highly effective]; and triphasic combined oral contraceptive pills)

  * Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Ability of a patient or a Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent document
* Body weight > 30 kg
* Must have a life expectancy of at least 12 weeks
* Cohort 1 (NSCLC cohort)

  * Ability to undergo a fresh tumor biopsy for the purpose of screening for this clinical trial (including able and willing to give valid written consent) to ability or to provide an available archival tumor sample taken less than 3 months prior to study enrollment (and not obtained prior to progression on a PD-1/PD-L1 inhibitor) if a fresh tumor biopsy is not feasible with an acceptable clinical risk; tumor lesions used for fresh biopsies should be the same lesions to be irradiated when possible and should not be the same lesions used as Response Evaluation Criteria in Solid Tumors (RECIST) target lesions, unless there are no other lesions accessible; additional, optional archival tumor tissue is also requested from before the prior PD-1 directed therapy
* Cohort 2 (colorectal cohort)

  * Ability to undergo a fresh tumor biopsy for the purpose of screening for this clinical trial (including able and willing to give valid written consent) to ability or to provide an available archival tumor sample taken less than 3 months prior to study enrollment if a fresh tumor biopsy is not feasible with an acceptable clinical risk; tumor lesions used for fresh biopsies should be the same lesions to be irradiated when possible and should not be the same lesions used as RECIST target lesions, unless there are no other lesions accessible
  * Microsatellite stable (MSS) tumor as documented by either:

    * Immunohistochemistry (IHC) testing that does not suggest loss of MLH-1, MSH-2, PMS2 or MSH6
    * Polymerase chain reaction (PCR) testing that does not suggest microsatellite instability (MSI)

Exclusion Criteria:

* Patients who have had systemic (chemotherapy, biologic therapy or radiotherapy) within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study
* Receipt of prior radiotherapy or condition for any reason that would contribute radiation dose that would exceed tolerance of normal tissues, at the discretion of the treating physician
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1)
* Patients who are receiving any other investigational agents
* Patients with untreated brain metastases, spinal cord compression, or leptomeningeal carcinomatosis should be excluded from this clinical trial; patients whose brain metastases have been treated may participate provided they show radiographic stability (defined as 2 brain images, both of which are obtained after treatment to the brain metastases; these imaging scans should both be obtained at least four weeks apart and show no evidence of intracranial progression); in addition, any neurologic symptoms that developed either as a result of the brain metastases or their treatment must have resolved or be stable either, without the use of steroids, or are stable on a steroid dose of =< 10 mg/day of prednisone or its equivalent (and anti-convulsants) for at least 14 days prior to the start of treatment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to tremelimumab and MEDI4736 or previous toxicity attributed to MEDI4736 or other PD-1 or PD-L1 directed therapy that led to drug discontinuation
* Prior exposure to immune-mediated therapy, including durvalumab and tremelimumab, except for anti-PD-1 or anti-PD-L1 therapy (including durvalumab) in NSCLC patients; this includes anti-CTLA-4 agents (prior treatment with these agents is NOT allowed in either cohort) and, excludes therapeutic anticancer vaccines, excluding therapeutic anticancer vaccines; exposure to other investigational agents may be permitted after discussion with the study principal investigator (PI)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because MEDI4736 (durvalumab), tremelimumab are immune checkpoint inhibitors with the potential for teratogenic or abortifacient effects, as is radiation therapy; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with MEDI4736(durvalumab), tremelimumab and radiation, breastfeeding should be discontinued if the mother is treated with MEDI4736(durvalumab), tremelimumab and radiation
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy or 180 days after the last dose of durvalumab + tremelimumab combination therapy, whichever is later
* Human immunodeficiency virus (HIV)-positive patients are ineligible; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Any concurrent chemotherapy, immune therapy, biologic, hormonal therapy for cancer treatment
* Current or prior use of immunosuppressive medication within 14 days before the first dose of their assigned IP; the following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra-articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
  * Steroids as pre-medication for hypersensitivity reactions (e.g., CT scan pre-medication)
* Major surgical procedure (as defined by the investigator) within 28 days prior to the first dose of IP; Note: local surgery of isolated lesions for palliative intent is acceptable
* History of allogeneic organ transplantation
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease, diverticulitis [with the exception of diverticulosis]; sarcoidosis syndrome, or other serious gastrointestinal [GI] chronic conditions associated with diarrhea; systemic lupus erythematosus; Wegener syndrome [granulomatosis with polyangiitis]; myasthenia gravis; Graves disease; rheumatoid arthritis; hypophysitis; uveitis, sarcoidosis syndrome, etc.) within the past 3 years prior to the start of treatment; the following are exceptions to this criterion:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement or psoriasis not requiring systemic treatment
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
  * Patients with celiac disease controlled by diet alone
* History of another primary malignancy except for

  * Malignancy treated with curative intent and with no known active disease >= 5 years before the first dose of study drug and of low potential risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease (e.g., cervical cancer in situ)
* Mean QT interval corrected for heart rate (QTc) >= 470 ms calculated from electrocardiograms (ECGs) using Fridericia's correction; abnormal ECGs should be repeated
* History of active primary immunodeficiency
* Known history of previous clinical diagnosis of tuberculosis
* Active infection including hepatitis B (known positive hepatitis B virus [HBV] surface antigen [HBsAg]) result or, hepatitis C; patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible; patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid (RNA); negative serologies documented over the past year are sufficient evidence of this
* Receipt of live, attenuated vaccine within 30 days prior to the first dose of investigational treatment; Note: patients, if enrolled, should not receive live vaccine during the study and up to 30 days after the last dose of investigational treatment
* Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational treatment or interpretation of patient safety or study results
* Any unresolved toxicity National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grade >= 2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

  * Patients with grade >= 2 neuropathy will be evaluated on a case-by-case basis after consultation with the study physician; patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the study physician
* Cohort 1 (NSCLC cohort)

  * In regards to administration of prior anti-PD-1 or anti PD-L1 antibodies, a patients:

    * Must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy
    * All adverse events (AEs) while receiving prior immunotherapy must have completely resolved or resolved to baseline prior to screening for this study
    * Must not have experienced a >= grade 3 immune related AE or an immune related neurologic or ocular AE of any grade while receiving prior immunotherapy; NOTE: subjects with endocrine AE of =< grade 2 are permitted to enroll if they are stably maintained on appropriate replacement therapy and are asymptomatic
    * Must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE, not have experienced recurrence of an AE if re-challenged, and not currently require maintenance doses of > 10 mg prednisone or equivalent per day
  * Eligibility for Food and Drug Administration (FDA)-approved agents targeting the EGFR, ROS1 or ALK pathway, which should be evaluated as per standard of care; exceptions to this requirement may be considered on a case-by-case basis by the principal investigator if the patient was previously treated with another targeted agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2026-01-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D Schoenfeld, Principal Investigator — Dana-Farber - Harvard Cancer Center LAO
Locations (42):
- United States (41):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Schoenfeld JD, Giobbie-Hurder A, Ranasinghe S, Kao KZ, Lako A, Tsuji J, Liu Y, Brennick RC, Gentzler RD, Lee C, Hubbard J, Arnold SM, Abbruzzese JL, Jabbour SK, Uboha NV, Stephans KL, Johnson JM, Park H, Villaruz LC, Sharon E, Streicher H, Ahmed MM, Lyon H, Cibuskis C, Lennon N, Jhaveri A, Yang L, Altreuter J, Gunasti L, Weirather JL, Mak RH, Awad MM, Rodig SJ, Chen HX, Wu CJ, Monjazeb AM, Hodi FS. Durvalumab plus tremelimumab alone or in combination with low-dose or hypofractionated radiotherapy in metastatic non-small-cell lung cancer refractory to previous PD(L)-1 therapy: an open-label, multicentre, randomised, phase 2 trial. Lancet Oncol. 2022 Feb;23(2):279-291. doi: 10.1016/S1470-2045(21)00658-6. Epub 2022 Jan 13. PMID 35033226

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 18 medical centers. The first participant was enrolled in August 2017 and the last in March 2019.
Pre-assignment Details: NSCLC: Ninety participants were randomized (30 per arm). A total of twelve participants either withdrew consent (N=5) before starting protocol therapy, were found to be ineligible (N=4), or progressed prior to starting protocol therapy (N=3) and were not included in the analysis.
  CRC: Twenty patients were randomized (10 per arm). One patient (Arm B) never started protocol therapy.
Groups:
- NSCLC Arm A (Tremelimumab, Durvalumab, HD-RT): Patients receive tremelimumab and durvalumab as in Arm C. Beginning at week 2, patients receive high dose radiation therapy QD over 10 days for up to 3 fractions.
  Durvalumab: Given IV
  Radiation Therapy: Undergo radiation therapy
  Tremelimumab: Given IV
- NSCLC Arm B (Tremelimumab, Durvalumab, LD-RT): Patients receive tremelimumab and durvalumab as in Arm C. Beginning at week 2, patients receive low dose radiation therapy every 6 hours BID on weeks 2, 6, 10 and 14.
  Durvalumab: Given IV
  Radiation Therapy: Undergo radiation therapy
  Tremelimumab: Given IV
- NSCLC Arm C (Tremelimumab, Durvalumab): Patients receive tremelimumab IV and durvalumab IV over 60 minutes every 4 weeks for up to 16 weeks in the absence of disease progression or unacceptable toxicity. Patients then receive durvalumab IV over 60 minutes 4 weeks after last combination dose for up to 9 additional doses.
  Durvalumab: Given IV
  Tremelimumab: Given IV
- CRC Arm A (Tremelimumab, Druvalumab, HD-RT): Patients receive tremelimumab IV and durvalumab IV over 60 minutes every 4 weeks for up to 16 weeks in the absence of disease progression or unacceptable toxicity. Patients then receive durvalumab IV over 60 minutes 4 weeks after last combination dose for up to 9 additional doses. Beginning at week 2, patients receive high dose radiation therapy QD over 10 days for up to 3 fractions.
  Durvalumab: Given IV
  Radiation Therapy: Undergo radiation therapy
  Tremelimumab: Given IV
- CRC Arm B (Tremelimumab, Dervalumab, LD-RT): Patients receive tremelimumab IV and durvalumab IV over 60 minutes every 4 weeks for up to 16 weeks in the absence of disease progression or unacceptable toxicity. Patients then receive durvalumab IV over 60 minutes 4 weeks after last combination dose for up to 9 additional doses. Beginning at week 2, patients receive low dose radiation therapy every 6 hours BID on weeks 2, 6, 10 and 14.
  Durvalumab: Given IV
  Radiation Therapy: Undergo radiation therapy
  Tremelimumab: Given IV
Period: Overall Study
Arm/Group | NSCLC Arm A (Tremelimumab, Durvalumab, HD-RT) | NSCLC Arm B (Tremelimumab, Durvalumab, LD-RT) | NSCLC Arm C (Tremelimumab, Durvalumab) | CRC Arm A (Tremelimumab, Druvalumab, HD-RT) | CRC Arm B (Tremelimumab, Dervalumab, LD-RT)
Started | 30 | 30 | 30 | 10 | 10
Received Protocol Therapy | 26 | 26 | 26 | 10 | 9
Completed | 26 | 26 | 26 | 10 | 9
Not Completed | 4 | 4 | 4 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 2 | 0 | 1
Not completed — Disease progression before treatment | 2 | 0 | 2 | 0 | 0
Not completed — Patient ineligible | 1 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants receiving at least one dose of protocol therapy.
Groups:
- CRC Arm A Tremelimumab, Durvalumab, HD-RT): Patients receive tremelimumab IV and durvalumab IV over 60 minutes every 4 weeks for up to 16 weeks in the absence of disease progression or unacceptable toxicity. Patients then receive durvalumab IV over 60 minutes 4 weeks after last combination dose for up to 9 additional doses.
  Beginning at week 2, patients receive high dose radiation therapy QD over 10 days for up to 3 fractions.
  Durvalumab: Given IV
  Radiation Therapy: Undergo radiation therapy
  Tremelimumab: Given IV
- CRC Arm B (Tremelimumab, Durvalumab, LD-RT): Patients receive tremelimumab IV and durvalumab IV over 60 minutes every 4 weeks for up to 16 weeks in the absence of disease progression or unacceptable toxicity. Patients then receive durvalumab IV over 60 minutes 4 weeks after last combination dose for up to 9 additional doses. Beginning at week 2, patients receive low dose radiation therapy every 6 hours BID on weeks 2, 6, 10 and 14..
  Durvalumab: Given IV
  Radiation Therapy: Undergo radiation therapy
  Tremelimumab: Given IV
- Total: Total of all reporting groups
Arm/Group | NSCLC Arm A (Tremelimumab, Durvalumab, HD-RT) | NSCLC Arm B (Tremelimumab, Durvalumab, LD-RT) | NSCLC Arm C (Tremelimumab, Durvalumab) | CRC Arm A Tremelimumab, Durvalumab, HD-RT) | CRC Arm B (Tremelimumab, Durvalumab, LD-RT) | Total
Number analyzed (Participants) | 26 | 26 | 26 | 10 | 9 | 97
Age, Continuous [Median (Full Range); unit: Years] | 65.5 [46.0 to 88.0] | 68.0 [45.0 to 77.0] | 65.5 [29.0 to 77.0] | 58 [38 to 79] | 59 [29 to 77] | 66.0 [29.0 to 88.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 9 | 6 | 5 | 39
  Male | 15 | 18 | 17 | 4 | 4 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 0 | 2 | 0 | 6
  Not Hispanic or Latino | 22 | 25 | 25 | 7 | 9 | 88
  Unknown or Not Reported | 1 | 0 | 1 | 1 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 1 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 3 | 0 | 3 | 8
  White | 22 | 22 | 21 | 7 | 6 | 78
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 1 | 3 | 0 | 7
Region of Enrollment [Number; unit: participants]
  United States | 26 | 26 | 26 | 10 | 9 | 97
ECOG Performance Status (PS) [Count of Participants; unit: Participants] — The Eastern Cooperative Oncology Group (ECOG) performance status (PS) scale measures a patient's functional status in relation to cancer. The scale describes a patient's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability. Scoring is as follows: 0 - Fully active; 1 - Restricted in strenuous activity; 2 - Restricted in work activity, but ambulatory and capable of self-care; 3 - Capable of limited self-care; 4 - Completely disabled; 5 - Dead.
  Participants
    0 (Fully active) | 6 | 9 | 5 | 6 | 5 | 31
    1 (Restricted in strenuous activities) | 19 | 17 | 20 | 4 | 4 | 64
    2 (Restricted in work; capable of self care) | 1 | 0 | 1 | 0 | 0 | 2
Histology [Count of Participants; unit: Participants]
  Adenocarcinoma | 16 | 21 | 19 | 10 | 9 | 75
  Squamous | 5 | 1 | 3 | 0 | 0 | 9
  Not specified | 5 | 4 | 4 | 0 | 0 | 13
Previous Radiotherapy [Count of Participants; unit: Participants]
  Yes | 16 | 17 | 20 | 2 | 3 | 58
  No | 10 | 9 | 6 | 8 | 6 | 39
Previous lines of therapy [Median (Inter-Quartile Range); unit: Lines of therapy] | 3 [2 to 4] | 3 [2 to 3] | 3 [2 to 4] | 4 [2 to 7] | 3 [1 to 7] | 3 [2 to 4]

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Determined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. NSCLC: The proportion of patients with response (complete response or partial response according to RECIST) will be compared for each pair-wise comparison of radiotherapy (RT)-containing therapy and control using chi- squared tests. The difference between the proportions responding will be presented with a 90% confidence interval. CRC: The proportion of patients with response will be presented with a 90% exact confidence interval.
Time Frame: Up to 2 years
Population: All patients receiving at least one regimen of protocol therapy.
Measure: Count of Participants; unit: Participants
Groups:
- NSCLC Arm A (Tremelimumab, Durvalumab, HD-RT): Patients receive tremelimumab and durvalumab as in Arm C. Beginning at week 2, patients receive high-dose radiation therapy QD over 10 days for up to 3 fractions.
  Durvalumab: Given IV
  Radiation Therapy: Undergo radiation therapy
  Tremelimumab: Given IV
- NSCLC Arm B (Tremelimumab, Durvalumab, LD-RT): Patients receive tremelimumab and durvalumab as in Arm C. Beginning at week 2, patients receive low-dose radiation therapy every 6 hours BID on weeks 2, 6, 10 and 14.
  Durvalumab: Given IV
  Radiation Therapy: Undergo radiation therapy
  Tremelimumab: Given IV
- CRC Arm A (Tremelimumab, Durvalumab, HD-RT): Patients receive tremelimumab IV and durvalumab IV over 60 minutes every 4 weeks for up to 16 weeks in the absence of disease progression or unacceptable toxicity. Patients then receive durvalumab IV over 60 minutes 4 weeks after last combination dose for up to 9 additional doses. Beginning at week 2, patients receive high-dose radiation therapy QD over 10 days for up to 3 fractions.
  Durvalumab: Given IV
  Radiation Therapy: Undergo radiation therapy
  Tremelimumab: Given IV
- CRC Arm B (Tremelimumab, Durvalumab, LD-RT): Patients receive tremelimumab IV and durvalumab IV over 60 minutes every 4 weeks for up to 16 weeks in the absence of disease progression or unacceptable toxicity. Patients then receive durvalumab IV over 60 minutes 4 weeks after last combination dose for up to 9 additional doses. Beginning at week 2, patients receive low-dose radiation therapy every 6 hours BID on weeks 2, 6, 10 and 14.
  Durvalumab: Given IV
  Radiation Therapy: Undergo radiation therapy
  Tremelimumab: Given IV
Arm/Group | NSCLC Arm A (Tremelimumab, Durvalumab, HD-RT) | NSCLC Arm B (Tremelimumab, Durvalumab, LD-RT) | NSCLC Arm C (Tremelimumab, Durvalumab) | CRC Arm A (Tremelimumab, Durvalumab, HD-RT) | CRC Arm B (Tremelimumab, Durvalumab, LD-RT)
Number analyzed (Participants) | 26 | 26 | 26 | 10 | 9
Participants | 3 | 2 | 3 | 0 | 0
Statistical Analysis 1: Comparison: NSCLC Arm A (Tremelimumab, Durvalumab, HD-RT) vs NSCLC Arm C (Tremelimumab, Durvalumab); Test type: Superiority; p = 0.99, Chi-squared; Difference between proportions = 0.0, 90% CI 2-sided [-14.6 to 14.6] — Arm A compared with Arm C; normal approximation for confidence interval
Statistical Analysis 2: Comparison: NSCLC Arm B (Tremelimumab, Durvalumab, LD-RT) vs NSCLC Arm C (Tremelimumab, Durvalumab); Test type: Superiority; p = 0.64, Chi-squared; Difference between proportions = -3.8, 90% CI 2-sided [-17.3 to 9.6] — Arm B compared with Arm C; normal approximation used for confidence interval

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Distributions are summarized using the Kaplan-Meier method. Median times for each therapy arm are accompanied by 90% confidence intervals based on log(-log(endpoint)) methodology. NSCLC: The pairwise comparisons between the durvalumab/tremelimumab alone and durvalumab/tremelimumab with RT arms will be conducted using Cox regression. CRC: No statistical comparisons conducted between Arms A and B.
Time Frame: From date of randomization until objective disease progression or death, whichever occurs first [up to 2 years]
Population: Patients receiving at least one regimen of protocol therapy.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | NSCLC Arm A (Tremelimumab, Durvalumab, HD-RT) | NSCLC Arm B (Tremelimumab, Durvalumab, LD-RT) | NSCLC Arm C (Tremelimumab, Durvalumab) | CRC Arm A (Tremelimumab, Durvalumab, HD-RT) | CRC Arm B (Tremelimumab, Durvalumab, LD-RT)
Number analyzed (Participants) | 26 | 26 | 26 | 10 | 9
Months | 4.0 [2.1 to 7.0] | 4.6 [2.1 to 7.2] | 3.3 [1.8 to 5.5] | 1.8 [1.5 to 2.0] | 1.6 [1.3 to 1.9]
Statistical Analysis 1: Comparison: NSCLC Arm A (Tremelimumab, Durvalumab, HD-RT) vs NSCLC Arm C (Tremelimumab, Durvalumab); Test type: Superiority; p = 0.92, Regression, Cox; Hazard Ratio (HR) = 0.81, 90% CI 2-sided [0.60 to 1.58]
Statistical Analysis 2: Comparison: NSCLC Arm B (Tremelimumab, Durvalumab, LD-RT) vs NSCLC Arm C (Tremelimumab, Durvalumab); Test type: Superiority; p = 0.55, Regression, Cox; Hazard Ratio (HR) = 0.83, 90% CI 2-sided [0.50 to 1.38]

3. Secondary Outcome: Overall Survival (OS)
Description: Distributions are summarized using the method of Kaplan-Meier. Median times for each therapy arm are accompanied by 90% confidence intervals based on log(-log(endpoint)) methodology. NSCLC: The pairwise comparisons between the durvalumab/tremelimumab alone and durvalumab/tremelimumab with RT arms are conducted using Cox regression. CRC: No statistical comparisons between arms were conducted.
Time Frame: From time of randomization to death from any cause [up to 2 years]
Population: Patients receiving at least one regimen of protocol therapy.
Measure: Median (90% Confidence Interval); unit: Months
Groups:
- Arm C (Tremelimumab, Durvalumab): Patients receive tremelimumab IV and durvalumab IV over 60 minutes every 4 weeks for up to 16 weeks in the absence of disease progression or unacceptable toxicity. Patients then receive durvalumab IV over 60 minutes 4 weeks after last combination dose for up to 9 additional doses.
  Durvalumab: Given IV
  Tremelimumab: Given IV
- CRC Arm A (Tremelimumab, Durvalumab, HD-RT): Patients receive tremelimumab IV and durvalumab IV over 60 minutes every 4 weeks for up to 16 weeks in the absence of disease progression or unacceptable toxicity. Patients then receive durvalumab IV over 60 minutes 4 weeks after last combination dose for up to 9 additional doses. Beginning at week 2, patients receive high dose radiation therapy QD over 10 days for up to 3 fractions.
  Durvalumab: Given IV
  Radiation Therapy: Undergo radiation therapy
  Tremelimumab: Given IV
- CRC Arm B (Tremelimumab, Durvalumab, LD-RT): Patients receive tremelimumab IV and durvalumab IV over 60 minutes every 4 weeks for up to 16 weeks in the absence of disease progression or unacceptable toxicity. Patients then receive durvalumab IV over 60 minutes 4 weeks after last combination dose for up to 9 additional doses. Beginning at week 2, patients receive low dose radiation therapy every 6 hours BID on weeks 2, 6, 10 and 14.
  Durvalumab: Given IV
  Radiation Therapy: Undergo radiation therapy
  Tremelimumab: Given IV
Arm/Group | NSCLC Arm A (Tremelimumab, Durvalumab, HD-RT) | NSCLC Arm B (Tremelimumab, Durvalumab, LD-RT) | Arm C (Tremelimumab, Durvalumab) | CRC Arm A (Tremelimumab, Durvalumab, HD-RT) | CRC Arm B (Tremelimumab, Durvalumab, LD-RT)
Number analyzed (Participants) | 26 | 26 | 26 | 10 | 9
Months | 9.7 [5.1 to NA] — The upper bound of the confidence interval was not reached | 9.1 [3.8 to 23.9] | NA [4.9 to NA] — The median OS and upper bound of the confidence interval were not reached. | 3.6 [2.2 to 6.4] | 4.2 [2.1 to 5.7]
Statistical Analysis 1: Comparison: NSCLC Arm B (Tremelimumab, Durvalumab, LD-RT) vs Arm C (Tremelimumab, Durvalumab); Test type: Superiority; p = 0.24, Regression, Cox; Hazard Ratio (HR) = 0.61, 90% CI 2-sided [0.30 to 1.22]
Statistical Analysis 2: Comparison: NSCLC Arm A (Tremelimumab, Durvalumab, HD-RT) vs Arm C (Tremelimumab, Durvalumab); Test type: Superiority; p = 0.44, Regression, Cox; Hazard Ratio (HR) = 0.72, 90% CI 2-sided [0.36 to 1.45]

4. Secondary Outcome: Objective Response Per Immune-related Response (irRC) Criteria
Description: NSCLC only: Proportions with irCR, irPR, irSD, irPD, and NA are presented with 90% exact binomial confidence intervals.
  The Immune-Related Response Criteria (irRC) is a set of published rules that defines when cancer tumors improve, stay the same, or worsen during treatment with an immuno-oncology drug. The response criteria are:
  irCR: Complete disappearance of all lesions, no new lesions, and confirmation by a repeat consecutive assessment no less than 4 weeks from date first documented; irPR: decrease in tumor burden >50% relative to baseline confirmed by repeat consecutive assessment at least 4 weeks later; irPD: increase in tumor burden >25% relative to nadir (minimum recorded tumor burden) confirmed by repeat consecutive assessment at least 4 weeks later; irSD: not meeting criteria for irCR or irPR in the absence of irPD.
Time Frame: Up to 2 years
Population: Patients receiving at least one regimen of protocol therapy.
Measure: Count of Participants; unit: Participants
Groups:
- Arm A (Tremelimumab, Durvalumab, HD-RT): Patients receive tremelimumab and durvalumab as in Arm C. Beginning at week 2, patients receive high dose radiation therapy QD over 10 days for up to 3 fractions.
  Durvalumab: Given IV
  Radiation Therapy: Undergo radiation therapy
  Tremelimumab: Given IV
- Arm B (Tremelimumab, Durvalumab, LD-RT): Patients receive tremelimumab and durvalumab as in Arm C. Beginning at week 2, patients receive low dose radiation therapy every 6 hours BID on weeks 2, 6, 10 and 14.
  Durvalumab: Given IV
  Radiation Therapy: Undergo radiation therapy
  Tremelimumab: Given IV
Arm/Group | Arm A (Tremelimumab, Durvalumab, HD-RT) | Arm B (Tremelimumab, Durvalumab, LD-RT) | Arm C (Tremelimumab, Durvalumab)
Number analyzed (Participants) | 26 | 26 | 26
Participants
  irCR | 0 | 0 | 0
  irPR | 3 | 2 | 2
  irSD | 9 | 11 | 9
  irPD | 9 | 8 | 11
  Missing/not available | 5 | 5 | 4

5. Secondary Outcome: Incidence of Grade 3-5 Adverse Events
Description: Assessed by Common Terminology Criteria for Adverse Events version 4.0. The proportions of subjects with grade-3 or higher adverse events (all attributions) are presented with 90% exact binomial confidence intervals.
Time Frame: Up to 2 years
Population: Participants who received at least one regimen of protocol therapy.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | NSCLC Arm A (Tremelimumab, Durvalumab, HD-RT) | NSCLC Arm B (Tremelimumab, Durvalumab, LD-RT) | NSCLC Arm C (Tremelimumab, Durvalumab) | CRC Arm A (Tremelimumab, Durvalumab, HD-RT) | CRC Arm B (Tremelimumab, Durvalumab, LD-RT)
Number analyzed (Participants) | 26 | 26 | 26 | 10 | 9
Percentage of participants | 11.5 [3 to 27] | 30.8 [16 to 49] | 15.4 [5 to 32] | 70.0 [39 to 91] | 77.8 [45 to 96]

6. Secondary Outcome: Local Control Rate and Abscopal Response Rate
Description: NSCLC: Local control - Having two or more scans with RECIST response of stable disease (SD), one response of SD followed by non-confirmed PR, or a confirmed response of PR.
  Abscopal response occurs when a local therapy, such as radiation therapy, not only shrinks the targeted tumor(s) but also leads to the shrinkage of untreated tumors elsewhere in the body. Abscopal response is measured using RECIST criteria (proportion of patients with complete (CR) or partial (PR) response to therapy).
Time Frame: Up to 2 years
Population: Participants receiving at least one regimen of protocol therapy.
Measure: Count of Participants; unit: Participants
Groups:
- Arm A (Tremelimumab, Durvalumab, HD-RT): Patients receive tremelimumab and durvalumab as in Arm C. Beginning at week 2, patients receive high-dose radiation therapy QD over 10 days for up to 3 fractions.
  Durvalumab: Given IV
  Radiation Therapy: Undergo radiation therapy
  Tremelimumab: Given IV
- Arm B (Tremelimumab, Durvalumab, LD-RT): Patients receive tremelimumab and durvalumab as in Arm C. Beginning at week 2, patients receive low-dose radiation therapy every 6 hours BID on weeks 2, 6, 10 and 14.
  Durvalumab: Given IV
  Radiation Therapy: Undergo radiation therapy
  Tremelimumab: Given IV
Arm/Group | Arm A (Tremelimumab, Durvalumab, HD-RT) | Arm B (Tremelimumab, Durvalumab, LD-RT) | Arm C (Tremelimumab, Durvalumab)
Number analyzed (Participants) | 26 | 26 | 26
Participants
  Local control | 9 | 6 | 8
  Abscopal response | 3 | 2 | 2

7. Secondary Outcome: Prognostic Effect of PD-L1 Expression
Description: NSCLC participants only: Pre-treatment levels of PD-L1 percent will be compared according to RECIST response using Wilcoxon rank-sum testing.
  PD-L1 percent: The percentage of tumor cells that positively express the PD-L1 protein (programmed cell death ligand 1). Tumors that express high amounts of PD-L1 (>50%) may respond well to checkpoint inhibitors (a type of immunotherapy drug).
Time Frame: Up to 2 years
Population: Participants in the NSCLC cohort with PD-L1 IHC evaluation. This analysis was pre-specified in the protocol to collect, analyze, and report data according to response and not by treatment Arm. Patients were classified into responders and non-responders according to RECIST criteria. PD-L1 percent was compared between these two groups of patients.
Measure: Mean (Standard Deviation); unit: Percent expression
Groups:
- Confirmed Responders: Participants with confirmed RECIST response of CR or PR.
- Non-responders: Participants without confirmed response of CR or PR.
Arm/Group | Confirmed Responders | Non-responders
Number analyzed (Participants) | 6 | 43
Percent expression | 15.8 (31.7) | 15.3 (25.2)
Statistical Analysis 1: Comparison: Confirmed Responders vs Non-responders; Test type: Superiority; p = 0.68, Wilcoxon (Mann-Whitney) — Unadjusted p-value

ADVERSE EVENTS:
Time Frame: Two years
Description: SAEs and non-SAE adverse events reflect all degrees of relatedness to study intervention.
  Non-SAE events are adverse events that were new or worsening relative to baseline.
  A 5% threshold was used for reporting non-SAE events (NSCLC: 4 or more of 78, CRC: 1 or more).
Arm/Group | NSCLC Arm A (Tremelimumab, Durvalumab, HD-RT) | NSCLC Arm B (Tremelimumab, Durvalumab, LD-RT) | NSCLC Arm C (Tremelimumab, Durvalumab) | CRC Arm A (Tremelimumab, Durvalumab, HD-RT) | CRC Arm B (Tremelimumab, Durvalumab, LD-RT)
All-Cause Mortality (participants affected / at risk) | 15/26 | 15/26 | 9/26 | 6/10 | 6/9
Serious Adverse Events (participants affected / at risk) | 9/26 | 11/26 | 8/26 | 5/10 | 6/9
Other Adverse Events (participants affected / at risk) | 25/26 | 24/26 | 24/26 | 9/10 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NSCLC Arm A (Tremelimumab, Durvalumab, HD-RT) (N=26) | NSCLC Arm B (Tremelimumab, Durvalumab, LD-RT) (N=26) | NSCLC Arm C (Tremelimumab, Durvalumab) (N=26) | CRC Arm A (Tremelimumab, Durvalumab, HD-RT) (N=10) | CRC Arm B (Tremelimumab, Durvalumab, LD-RT) (N=9)
Anemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cyanosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (4)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Edema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hepatic Failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Encephalitis infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip/spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Alkaline Phosphatase Increased (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Bilirubin Increased (Investigations) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Death - Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Death - Metastatic primary lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastatic Disease To The Brain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Bronchial Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 4 (4) | 1 (2) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Death - Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Maculo-papular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral Ischemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Superior Vena Cava Syndrome (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NSCLC Arm A (Tremelimumab, Durvalumab, HD-RT) (N=26) | NSCLC Arm B (Tremelimumab, Durvalumab, LD-RT) (N=26) | NSCLC Arm C (Tremelimumab, Durvalumab) (N=26) | CRC Arm A (Tremelimumab, Durvalumab, HD-RT) (N=10) | CRC Arm B (Tremelimumab, Durvalumab, LD-RT) (N=9)
Absolute Neutrophil Count (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 4 (6) | 7 (13) | 4 (7) | 4 (5) | 6 (15)
Decreased Hematocrit (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (6)
Decreased MCHC (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (3)
Decreased RBC (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Elevated Absolute Monocyte (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Elevated Bands (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Elevated BUN (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eosinophil Count Elevated (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased Monocyte Count (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased Neutrophils (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Increased Platelets (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased RDW (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Monocyte Count Increased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sinus Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 4 (7)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 3 (5) | 1 (2) | 3 (20) | 3 (4) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (4)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 2 (10)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (4) | 4 (7) | 5 (12) | 0 (0) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 6 (10) | 7 (15) | 7 (20) | 5 (10) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Fecal Incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 7 (9) | 7 (12) | 5 (12) | 3 (4)
Oral Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (9) | 3 (6) | 0 (0) | 4 (8) | 3 (4)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Edema Limbs (General disorders) | 2 (2) | 2 (2) | 3 (5) | 4 (5) | 2 (4)
Fatigue (General disorders) | 11 (22) | 11 (21) | 9 (37) | 6 (12) | 5 (9)
Fever (General disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 2 (2)
Flu Like Symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gait Disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 2 (5) | 2 (2) | 0 (0) | 2 (2)
Opioid Overdose (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 4 (11) | 3 (6) | 2 (4) | 1 (1) | 0 (0)
Cytokine Release Syndrome (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 2 (4) | 1 (5) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (4) | 2 (2) | 2 (4) | 1 (1) | 0 (0)
Pigtail Cath Malfunction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wrist Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Alanine Aminotransferase Increased (Investigations) | 2 (12) | 1 (1) | 2 (3) | 1 (1) | 1 (1)
Alkaline Phosphatase Increased (Investigations) | 7 (18) | 3 (4) | 6 (9) | 3 (4) | 4 (5)
ALT Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amylase Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 2 (9) | 2 (2) | 1 (1) | 3 (4) | 6 (7)
Blood Bilirubin Increased (Investigations) | 2 (3) | 1 (2) | 1 (1) | 1 (1) | 2 (3)
Creatinine Increased (Investigations) | 3 (15) | 3 (3) | 3 (14) | 1 (1) | 1 (1)
Decreased ALT (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Decreased Amylase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased BUN (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased Carbon Dioxide (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Decreased Chloride (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Decreased GFR (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased Hematocrit (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (5)
Decreased Lipase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Decreased MCH (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Decreased MCHC (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (3)
Decreased MCV (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased Protein (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased RBC (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Decreased Total Protein (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Decreased Urea Nitrogen (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Elevated Ammonia (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Elevated Bands (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Elevated Carbon Dioxide (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Elevated Lactic Acid (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Elevated RDW (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Elevated WBC (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GGT Increased (Investigations) | 6 (9) | 3 (3) | 0 (0) | 3 (4) | 4 (4)
Increased ANC (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Increased BUN (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased GFR (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased Monocytes (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Increased Neutrophil (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased Prothrombin Time (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Increased RDW (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Increased Red Cell Distribution Width (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased Total Protein (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Increased WBC (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased White Blood Cells (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INR Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
LDH Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte Count Decreased (Investigations) | 4 (8) | 2 (4) | 4 (10) | 3 (7) | 6 (14)
Monocyte Count Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Phosphorus Elevated (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet Count Decreased (Investigations) | 1 (1) | 1 (1) | 2 (2) | 1 (2) | 1 (1)
PT Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serum Amylase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight Loss (Investigations) | 3 (3) | 3 (3) | 2 (5) | 1 (3) | 1 (2)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 5 (9) | 8 (18) | 9 (15) | 6 (10) | 3 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (4) | 2 (4) | 1 (1) | 3 (5) | 1 (1)
Failure To Thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 3 (9) | 6 (7) | 3 (7)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 4 (12) | 0 (0) | 1 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (9) | 3 (3) | 5 (8) | 4 (9) | 4 (7)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 3 (4)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (11) | 2 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (5) | 0 (0) | 1 (1) | 2 (5) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4) | 3 (7) | 4 (8) | 5 (15) | 4 (10)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 2 (3) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 4 (10) | 2 (8) | 4 (7) | 1 (1)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (3)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 2 (3) | 1 (4) | 1 (1)
Joint Range Of Motion Decreased Lumbar Spine (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle Weakness Right-Sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (17) | 1 (1) | 2 (6) | 1 (1) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (8) | 2 (3) | 0 (0) | 0 (0)
Abducens Nerve Disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 5 (9) | 2 (3) | 1 (4) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 1 (3) | 4 (10) | 3 (9) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 (0) | 2 (6) | 3 (17) | 1 (1) | 2 (3)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (6) | 4 (9) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (14) | 2 (2) | 1 (1) | 0 (0) | 1 (2)
Insomnia (Psychiatric disorders) | 2 (4) | 1 (3) | 4 (8) | 2 (5) | 2 (3)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Increased Urine Urobilinogen (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Urine Discoloration (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal Hemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (8) | 4 (9) | 5 (16) | 2 (3) | 1 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (9) | 4 (7) | 9 (18) | 3 (4) | 4 (8)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 3 (5) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (4) | 1 (1) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 2 (11) | 1 (2) | 2 (9) | 2 (5) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (43) | 5 (9) | 3 (17) | 1 (2) | 0 (0)
Rash Acneiform (Skin and subcutaneous tissue disorders) | 1 (4) | 1 (2) | 3 (12) | 0 (0) | 0 (0)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 7 (28) | 3 (8) | 5 (8) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypotension (Vascular disorders) | 3 (3) | 1 (1) | 2 (2) | 1 (3) | 3 (5)
Thromboembolic Event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-30): https://cdn.clinicaltrials.gov/large-docs/43/NCT02888743/Prot_SAP_000.pdf